CLINICAL TRIAL: NCT01667471
Title: Long-term, Interventional, Open Label Extension Study Evaluating the Safety of Tocilizumab Treatment in Patients With Polyarticular-course Juvenile Idiopathic Arthritis Who Completed the Global, Multinational Trial (WA19977)
Brief Title: A Long-Term Extension Study of RoActemra/Actemra (Tocilizumab) in Patients With Juvenile Idiopathic Arthritis Who Completed WA19977 Core Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25756; 2011-001097-25 (EudraCT Number)
Record Dates: First submitted 2012-08-15; First posted 2012-08-17 (Estimated); Results first posted 2015-10-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — tocilizumab

ARMS (1):
- RoActemra/Actemra (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 8 mg/kg iv every 4 weeks, 104 weeks

SUMMARY:
This long-term, open-label extension study will evaluate the safety of RoActemra/Actemra (tocilizumab) in patients with polyarticular-course juvenile idiopathic arthritis who completed the WA19977 core study. Patients aged 9-18 years with at least JIA ACR30 clinical response to RoActemra/Actemra in the core study will be eligible to receive RoActemra/Actemra 8 mg/kg intravenously every 4 weeks. Anticipated time on study treatment is 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients 9 to 18 years of age who completed visit 33 (week 104) of WA19977 study with at least JIA ACR30 clinical response to RoActemra/Actemra relative to baseline in WA19977, with no AEs, SAEs or conditions that lead to unacceptable risk of continued treatment
* Scheduled to receive first RoActemra/Actemra infusion in this study between 4 and 6 weeks after the last IV infusion in the core study
* Females of child-bearing potential and males with female partners of child-bearing potential must agree to use effective contraception as defined by protocol

Exclusion Criteria:

* Patients with, according to investigator judgment, not satisfactory benefit from RoActemra/Actemra therapy within WA19977
* Treatment with any investigational agent since the last administration of study drug in the core study WA19977 or current participation in another clinical trial except WA19977
* Patient developed any other autoimmune rheumatic disease or overlap syndrome other than the permitted polyarticular-course JIA subsets: rheumatoid factor positive or negative JIA or extended oligoarticular JIA
* Patient is pregnant , lactating, or intending to become pregnant during the study and up to 12 weeks after the last administration of study drug
* Any significant concomitant disease or medical or surgical condition
* History of significant allergic or infusion reactions to prior biologic therapy
* Known current active acute, subacute, chronic or history of recurrent infection; patients suffering from ongoing active infections with Epstein Barr virus, herpes zoster or recurrent history of urinary tract infection can be included after the (acute) infection has been excluded or subsided
* Positive for latent tuberculosis (TB)
* Currently active asthma for which the patient has required the use of oral or parenteral corticosteroids for >/= 2 weeks within 6 months prior to entering the study
* Inadequate hepatic, renal or bone marrow function

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2012-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Germany (3):
  - Bremen
  - Frankfurt am Main
  - Sankt Augustin

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab 8 mg/kg: Participants received tocilizumab 8 mg/kg intravenously (IV) every 4 weeks up to 104 weeks or until tocilizumab was commercially available for polyarticular-course Juvenile Idiopathic Arthritis (pcJIA).
Period: Overall Study
Arm/Group | Tocilizumab 8 mg/kg
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug were included in the Safety Analysis Set.
Groups:
- Tocilizumab 8 mg/kg: Participants received tocilizumab 8 mg/kg IV every 4 weeks up to 104 weeks or until tocilizumab was commercially available for pcJIA.
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.4 (3.2)
Gender [Count of Participants; unit: Participants]
  Female | 6
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events of Special Interest and Study-Drug Related Adverse Events
Description: Adverse Events (AEs) and Serious Adverse Events (SAEs) were recorded from the first day of tocilizumab administration until 4 weeks after administration of the last dose of tocilizumab. AEs of special interest were Infections (including all opportunistic infections and non-serious infections as defined by those treated with IV anti-infectives), Myocardial infarction/Acute coronary syndrome, Gastrointestinal perforations and related events, Malignancies, Anaphylaxis/Hypersensitivity reactions, Demyelinating disorders, Stroke. Bleeding events, Hepatic events and Macrophage activation syndrome (MAS).
Time Frame: Baseline and every 4 weeks up to Week 76 and Final Follow-Up Visit (up to 82 weeks)
Population: Safety Analysis Set
Measure: Number; unit: participants
Groups:
- Tocilizumab: Participants received tocilizumab 8 mg/kg IV every 4 weeks up to 104 weeks or until tocilizumab was commercially available for pcJIA.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 7
participants
  Drug related AEs | 6
  Drug related SAEs | 0
  AEs of special interest | 1
  Drug-related AEs of special interest | 1

2. Secondary Outcome: Percentage of Participants With Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) 30/50/70/90 by Visit
Description: The six JIA ACR components comprised of: 1) Physician's global assessment of disease activity, 2) Parent/Participant's global assessment of overall well-being, 3) Maximum number of joints with active arthritis, 4) Number of joints with limitation of movement, 5) Erythrocyte Sedimentation Rate (ESR) and/or C-reactive Protein (CRP), and 6) Childhood Health Assessment Questionnaire - Disease Index (CHAQ-DI).
  At an assessment visit, a JIA ACR30/50/70/90 response in comparison to Baseline was defined as: At least three of the six JIA ACR core components improving by at least 30 percent (%), 50%, 70%, or 90% respectively and no more than one of the remaining JIA ACR core components worsening by more than 30%.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 60, 72 and Final Follow-Up Visit (up to 82 weeks)
Population: Safety Analysis Set; number (n) = number of participants analyzed for the given parameter at the specified visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 7
percentage of participants
  Baseline JIA ACR30 (n=7) | 85.7
  Week 12 JIA ACR30 (n=7) | 100.0
  Week 24 JIA ACR30 (n=7) | 100.0
  Week 36 JIA ACR30 (n=7) | 100.0
  Week 48 JIA ACR30 (n=6) | 100.0
  Week 60 JIA ACR30 (n=6) | 100.0
  Week 72 JIA ACR30 (n=2) | 100.0
  Follow-Up JIA ACR30 (n=7) | 100.0
  Baseline JIA ACR50 (n=7) | 85.7
  Week 12 JIA ACR50 (n=7) | 100.0
  Week 24 JIA ACR50 (n=7) | 100.0
  Week 36 JIA ACR50 (n=7) | 100.0
  Week 48 JIA ACR50 (n=6) | 100.0
  Week 60 JIA ACR50 (n=6) | 100.0
  Week 72 JIA ACR50 (n=2) | 100.0
  Follow-Up JIA ACR50 (n=7) | 100.0
  Baseline JIA ACR70 (n=6) | 85.7
  Week 12 JIA ACR70 (n=7) | 100.0
  Week 24 JIA ACR70 (n=7) | 100.0
  Week 36 JIA ACR70 (n=7) | 100.0
  Week 48 JIA ACR70 (n=6) | 100.0
  Week 60 JIA ACR70 (n=6) | 100.0
  Week 72 JIA ACR70 (n=2) | 100.0
  Follow-Up JIA ACR70 (n=7) | 100.0
  Baseline JIA ACR90 (n=6) | 85.7
  Week 12 JIA ACR90 (n=7) | 85.7
  Week 24 JIA ACR90 (n=7) | 57.1
  Week 36 JIA ACR90 (n=7) | 71.4
  Week 48 JIA ACR90 (n=6) | 83.3
  Week 60 JIA ACR90 (n=6) | 66.7
  Week 72 JIA ACR90 (n=2) | 100.0
  Follow-Up JIA ACR90 (n=7) | 85.7

3. Primary Outcome: Number of AEs of Special Interest and Study Drug Related AEs
Description: AEs and SAEs were recorded from the first day of tocilizumab administration until 4 weeks after administration of the last dose of tocilizumab.
Time Frame: Baseline and every 4 weeks up to Week 76 and Final Follow-Up Visit (up to 82 weeks)
Population: Safety Analysis Set
Measure: Number; unit: adverse events
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 7
adverse events
  Drug related AEs | 22
  Drug related SAEs | 0
  AEs of special interest | 2
  Drug-related AEs of special interest | 2

4. Secondary Outcome: Percentage of Participants With Inactive Disease by Visit
Description: A participant was defined to show inactive disease if all of the following criteria were applied: 1) No joints with active arthritis (no joints with swelling and no joints with lack of motion), 2) No fever, rash, serositis, splenomegaly, or generalized lymphadenopathy attributable to JIA, 3) No active uveitis, 4) ESR and/or CRP within normal range, and 5) Physician's global assessment of disease activity equals (=) 0 millimeters (mm) on a Visual analog scale (VAS).
Time Frame: Baseline, Weeks 12, 24, 36, 48, 60, 72 and Final Follow-Up Visit (up to 82 weeks)
Population: Safety Analysis Set; n = number of participants analyzed for the given parameter at the specified visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 7
percentage of participants
  Baseline(n=7) | 57.1
  Week 12 (n=7) | 42.9
  Week 24 (n=7) | 14.3
  Week 36 (n=7) | 42.9
  Week 48 (n=6) | 16.7
  Week 60 (n=6) | 33.3
  Week 72 (n=2) | 50.0
  Follow-Up (n=7) | 57.1

5. Secondary Outcome: Percentage of Participants Achieving Clinical Remission (CR) at Each Visit
Description: CR was defined as "clinical remission with medication (CRem)". A participant was in CR if inactive disease was observed for a minimum of 6 consecutive months.
Time Frame: Baseline, Screening, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76 and Final Follow-Up Visit (up to 82 weeks)
Population: Safety Analysis Set; n = number of participants analyzed for the given parameter at the specified visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 7
percentage of participants
  Baseline (n=7) | 0.0
  Screening (n=7) | 0.0
  Week 4 (n=7) | 0.0
  Week 8 (n=7) | 0.0
  Week 12 (n=7) | 0.0
  Week 16 (n=7) | 0.0
  Week 20 (n=7) | 0.0
  Week 24 (n=7) | 0.0
  Week 28 (n=7) | 14.3
  Week 32 (n=7) | 14.3
  Week 36 (n=7) | 14.3
  Week 40 (n=6) | 16.7
  Week 44 (n=6) | 16.7
  Week 48 (n=6) | 16.7
  Week 52 (n=6) | 16.7
  Week 56 (n=6) | 16.7
  Week 60 (n=6) | 0.0
  Week 64 (n=5) | 0.0
  Week 68 (n=3) | 0.0
  Week 72 (n=2) | 0.0
  Week 76 (n=1) | 0.0
  Follow-Up (n=7) | 0.0

6. Secondary Outcome: Physicians Assessment of Global Activity (VAS)
Description: The participant's treating physician provided a rating of the participant's arthritis disease activity on a 0 to 100 mm horizontal scale. The extreme left end of the line, score 0 represented 'arthritis inactive' (ie, symptom-free and no arthritis symptoms) and the extreme right end score 100 represented 'arthritis very active'. A higher score indicated more disease activity.
Time Frame: Baseline, Weeks 12, 24, 28, 32, 36, 48, 60, 72 and Final Follow-Up Visit (up to 82 weeks)
Population: Safety Analysis Set; n = number of participants analyzed at the specified visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 7
mm
  Baseline (n=7) | 12.0 (30.4)
  Week 12 (n=7) | 2.3 (2.9)
  Week 24 (n=7) | 5.4 (6.1)
  Week 28 (n=1) | 1.0 (0.0)
  Week 32 (n=2) | 29.0 (8.5)
  Week 36 (n=7) | 5.0 (7.9)
  Week 48 (n=6) | 5.7 (8.2)
  Week 60 (n=6) | 5.7 (8.7)
  Week 72 (n=2) | 1.0 (1.4)
  Follow-Up (n=7) | 5.0 (8.7)

7. Secondary Outcome: Parent or Participant's Assessment of Global Activity (VAS)
Description: The participant or parent/guardian, as appropriate, provided a rating of the participant's well-being on a 0 to 100 mm horizontal scale. The extreme left end of the line Score 0 represented 'very well' (ie, symptom-free and no arthritis disease activity) and the extreme right end score 100 represented 'very poor' (ie, maximum arthritis disease activity). A higher score indicated poorer well-being.
Time Frame: Baseline, Weeks 12, 24, 28, 32, 36, 48, 60, 72 and Final Follow-Up Visit (up to 82 weeks)
Population: Safety Analysis Set; n = number of participants analyzed at the specified visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 7
mm
  Baseline (n=7) | 10.1 (20.0)
  Week 12 (n=7) | 7.1 (8.1)
  Week 24 (n=7) | 16.4 (19.9)
  Week 28 (n=1) | 1.0 (0.0)
  Week 32 (n=2) | 22.5 (24.7)
  Week 36 (n=7) | 12.1 (18.4)
  Week 48 (n=6) | 11.7 (13.9)
  Week 60 (n=6) | 10.2 (13.8)
  Week 72 (n=2) | 3.5 (4.9)
  Follow-Up (n=7) | 9.7 (16.0)

8. Secondary Outcome: Number of Joints With Active Arthritis
Description: Joints with active arthritis were defined as joints with swelling or pain and limited of motion. The maximum number of joints with active arthritis was 71.The joint assessment was performed by an independent assessor who was not the treating physician and who was blinded to all other aspects of the participant's efficacy and safety data.
Time Frame: Baseline, Weeks 12, 24, 28, 32, 36, 48, 60, 72 and Final Follow-Up Visit (up to 82 weeks)
Population: Safety Analysis Set; n = number of participants analyzed at the specified visit.
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 7
joints
  Baseline (n=7) | 0.9 (2.3)
  Week 12 (n=7) | 0.3 (0.8)
  Week 24 (n=7) | 1.0 (2.6)
  Week 28 (n=1) | 1.0 (0.0)
  Week 32 (n=2) | 1.5 (0.7)
  Week 36 (n=7) | 1.1 (2.2)
  Week 48 (n=6) | 0.0 (0.0)
  Week 60 (n=6) | 0.3 (0.8)
  Week 72 (n=2) | 0.0 (0.0)
  Follow-Up (n=7) | 0.3 (0.8)

9. Secondary Outcome: Number of Joints With Lack of Motion
Description: Joints with lack of movement were assessed. The maximum number of joints with lack of movement was 67. The joint assessment was performed by an independent assessor who was not the treating physician and who was blinded to all other aspects of the participant's efficacy and safety data.
Time Frame: Baseline, Weeks 12, 24, 28, 32, 36, 48, 60, 72 and Final Follow-Up Visit (up to 82 weeks)
Population: Safety Analysis Set; n = number of participants analyzed at the specified visit.
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 7
joints
  Baseline (n=7) | 1.4 (2.7)
  Week 12 (n=7) | 2.6 (5.1)
  Week 24 (n=7) | 2.4 (3.2)
  Week 28 (n=1) | 1.0 (0.0)
  Week 32 (n=2) | 5.5 (7.8)
  Week 36 (n=7) | 1.7 (2.4)
  Week 48 (n=6) | 2.7 (5.2)
  Week 60 (n=6) | 1.8 (3.0)
  Week 72 (n=2) | 0.0 (0.0)
  Follow-Up (n=7) | 2.9 (4.8)

10. Secondary Outcome: Erythrocyte Sedimentation Rate
Description: ESR is a marker of inflammation and was measured as millimeters per hour (mm/h). Healthy individuals have low ESR. Higher ESR indicate inflammation.
Time Frame: Baseline, Weeks 4, 8,12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76 and Final Follow-Up Visit (up to 82 weeks)
Population: Safety Analysis Set; n = number of participants analyzed at the specified visit.
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 7
mm/h
  Baseline (n=7) | 4.9 (5.1)
  Week 4 (n=7) | 3.0 (1.9)
  Week 8 (n=7) | 2.9 (2.3)
  Week 12 (n=7) | 3.0 (2.0)
  Week 16 (n=7) | 8.6 (16.1)
  Week 20 (n=7) | 2.6 (0.8)
  Week 24 (n=7) | 2.7 (1.4)
  Week 28 (n=5) | 3.4 (3.1)
  Week 32 (n=7) | 4.3 (4.2)
  Week 36 (n=7) | 4.3 (2.5)
  Week 40 (n=6) | 2.0 (1.8)
  Week 44 (n=6) | 2.7 (1.5)
  Week 48 (n=6) | 3.8 (1.5)
  Week 52 (n=6) | 3.2 (3.6)
  Week 56 (n=6) | 2.3 (1.6)
  Week 60 (n=6) | 10.2 (12.7)
  Week 64 (n=5) | 3.2 (2.4)
  Week 68 (n=3) | 10.0 (7.2)
  Week 72 (n=2) | 4.5 (0.7)
  Week 76 (n=1) | 2.0 (0.0)
  Follow-Up (n=7) | 4.3 (2.8)

11. Secondary Outcome: CHAQ-DI Score
Description: The CHAQ-DI questionnaire consisted of 30 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities. Each domain had at least two component questions and if applicable to the participant there were four possible responses (0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, 3 = unable to do). The CHAQ-DI score is the sum of the domain scores divided by the number of domains that have a non-missing score. This overall score ranges from 0 (best) to 3 (worst).
Time Frame: Baseline, Weeks 12, 24, 28, 32, 36, 48, 60, 72, and Final Follow-Up Visit (up to 82 weeks)
Population: Safety Analysis Set; n = number of participants analyzed at the specified visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 7
score on a scale
  Baseline (n=7) | 0.0 (0.0)
  Week 12 (n=7) | 0.04 (0.09)
  Week 24 (n=7) | 0.14 (0.20)
  Week 28 (n=1) | 0.00 (0.0)
  Week 32 (n=2) | 0.19 (0.27)
  Week 36 (n=7) | 0.13 (0.33)
  Week 48 (n=6) | 0.00 (0.00)
  Week 60 (n=6) | 0.21 (0.51)
  Week 72 (n=2) | 0.00 (0.00)
  Follow-Up (n=7) | 0.00 (0.00)

12. Secondary Outcome: Parent or Participant's Assessment of Pain (VAS)
Description: Parents or participants rated participant's pain by placing a horizontal line on a VAS of 0 (no pain)- 100 mm (severe pain).
Time Frame: Baseline, Weeks 12, 24, 28, 32, 36, 48, 60, 72, and Final Follow-Up Visit (up to 82 weeks)
Population: Safety Analysis Set; n = number of participants analyzed at the specified visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 7
mm
  Baseline (n=7) | 10.9 (21.8)
  Week 12 (n=7) | 7.0 (10.0)
  Week 24 (n=7) | 13.7 (16.7)
  Week 28 (n=1) | 1.0 (0.0)
  Week 32 (n=2) | 28.5 (17.7)
  Week 36 (n=7) | 10.6 (15.9)
  Week 48 (n=6) | 12.3 (13.6)
  Week 60 (n=6) | 10.2 (13.8)
  Week 72 (n=2) | 4.0 (5.7)
  Follow-Up (n=7) | 9.9 (15.9)

13. Secondary Outcome: CRP Levels
Description: CRP an acute phase protein, is a marker of inflammation. CRP was measured as milligrams per deciliter (mg/dL).
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76 and Final Follow-Up Follow-Up Visit (up to 82 weeks)
Population: Safety Analysis Set; n = number of participants analyzed at the specified visit.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 7
mg/dL
  Baseline (n=7) | 0.03 (0.01)
  Week 4 (n=7) | 0.05 (0.07)
  Week 8 (n=7) | 0.02 (0.02)
  Week 12 (n=7) | 0.03 (0.01)
  Week 16 (n=7) | 0.23 (0.54)
  Week 20 (n=7) | 0.05 (0.07)
  Week 24 (n=7) | 0.03 (0.02)
  Week 28 (n=6) | 0.02 (0.02)
  Week 32 (n=7) | 0.03 (0.02)
  Week 36 (n=7) | 0.02 (0.02)
  Week 40 (n=6) | 0.03 (0.02)
  Week 44 (n=6) | 0.03 (0.02)
  Week 48 (n=6) | 0.03 (0.02)
  Week 52 (n=6) | 0.02 (0.02)
  Week 56 (n=6) | 0.03 (0.02)
  Week 60 (n=6) | 0.38 (0.90)
  Week 64 (n=5) | 0.03 (0.03)
  Week 68 (n=3) | 0.09 (0.10)
  Week 72 (n=2) | 0.04 (0.04)
  Week 76 (n=1) | 0.05 (0.0)
  Follow-Up (n=7) | 0.05 (0.06)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the date of screening until the final Follow-Up Visit (up to 82 weeks).
Arm/Group | Tocilizumab 8 mg/kg
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab 8 mg/kg (N=7)
Appendicitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab 8 mg/kg (N=7)
Neutropenia (Blood and lymphatic system disorders) | 1
Aortic valve incompetence (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Epigastric discomfort (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Injection site swelling (General disorders) | 1
Local swelling (General disorders) | 1
Vaccination site reaction (General disorders) | 1
Acute tonsillitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 4
Herpes simplex (Infections and infestations) | 1
Lice infestation (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Scarlet fever (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 3
Vulvovaginal mycotic infection (Infections and infestations) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Biopsy kidney (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Foot deformity (Musculoskeletal and connective tissue disorders) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.